CLINICAL TRIAL: NCT03113552
Title: Prognostic Impact of the Location of Mitral Valve Prolapse on the Long-term Results of Mitral Plasty
Acronym: IPPVM
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2013_843_0002
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-02

CONDITIONS: Mitral Valve Prolapse; Mitral Plasty
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mitral insufficiency (MI) accounts for 24% of adult valvulopathies and affects 7% of subjects older than 75 years. They are the second leading cause of valvulopathy in Europe. The most common etiology is the associated valvular prolapse. Mitral surgery remains the reference treatment for symptomatic MI. The success of this procedure depends on the mitral valve geometry and the location of the prolapse. The site of the prolapse, whether monovalvular, localized to the posterior or anterior leaflet, or bivalvular, influences the possibilities and probably the long-term results of the plasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated between 1988 and 2011
* Presence of a valvular prolapse diagnosed by echocardiography
* Possibility of a complete clinical evaluation at the time of the initial echocardiography

Exclusion Criteria:

* Ischemic MI (including papillary muscle rupture)
* Presence of significant aortic valvulopathy, mitral valvular stenosis or congenital disease
* History of cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study of the long-term survival of patients who have had mitral valve prolapse for mitral valve prolapse in Amiens according to the location of the prolapse
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2013-02-04 (Actual); Primary Completion 2028-07-04 (Estimated); Study Completion 2028-07-04 (Estimated)

PRIMARY OUTCOMES:
Survival defines as the time between the date of surgery and the death or date of the last news | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France